CLINICAL TRIAL: NCT06868498
Title: Train and EMPOWER A Community Health Workforce to Achieve Equity and Reduce Disparities in Mental Health
Acronym: TEACH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0042.3; 1U01MD019540-01 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: CHW Certification
Keywords: CHW certification; Undergraduate students; University of Texas at Arlington; Baylor Scott &amp; White; Social Work; Community Health Worker; EMPOWER Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMPOWER-trained CHWs (Experimental): Undergraduate students at the University of Texas at Arlington will engage in a semester-long course for training of students as CHWs with additional EMPOWER training for delivering a brief trans-diagnostic psychosocial intervention. CHW certified students will then engage in an internship at Baylor Scott and White Health.
  Interventions: Other: A semester-long course for training of students as CHWs with additional EMPOWER training for delivering a brief trans-diagnostic psychosocial intervention.
- Non-EMPOWER-trained interns (No Intervention): Intern health workers who have not undergone the EMPOWER training curriculum will engage in an internship at Baylor Scott and White Health.

INTERVENTIONS:
Other: A semester-long course for training of students as CHWs with additional EMPOWER training for delivering a brief trans-diagnostic psychosocial intervention. — Students will participate in a special topics course resulting in a CHW certification with the state of Texas. The course will focus on behavioral activation interventions. Undergraduate Bachelor of Social Work (BSWs) students will then be deployed to the health system as certified CHWs with mental health training to provide a sufficient level of care for many, and an entry point to clinical care for those who have needs that are currently unaddressed.
  Arms: EMPOWER-trained CHWs

SUMMARY:
The investigators suggest a multi-step approach to improve access to mental health care for minority groups. The plan focuses on three goals: increasing diversity in the mental health workforce, bringing more expertise into the community, and strengthening the community's ability to address the factors that impact mental health.

To do this, the TEACH study team will work with students from underrepresented racial and ethnic groups at a minority-serving school. Students will be provided the opportunity to obtain their CHW Certification while receiving course credit for their degree. Students will then be eligible to participate in an internship to utilize their skills. The TEACH study team will help these students with their training, supervision, and ongoing support. These students will then be able to work with their communities to tackle common mental health issues and the social factors that contribute to those problems.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled as a UTA undergraduate student with unmet internship hours
* Must be aged 18 and over
* Must be able to provide informed consent.
* Must have successful completion of the UTA CHW/EMPOWER course (Phase 2) and/or State of Texas CHW certification (for non-EMPOWER-trained CHWs) at the start of internship

Exclusion Criteria:

* Under 18 years
* Not enrolled as an undergraduate student at UTA
* Unable to provide informed consent
* Non-successful completion of EMPOWER course and/or State of Texas CHW certification at the start of internship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Job Placement | 12 months after the intervention has ended
  Data collected regarding career placement and/or further educational pursuits (i.e. MSW)

SECONDARY OUTCOMES:
Depression | Baseline, an average of 5 months after the start of the intervention, and immediately after the intervention, an average of 10 months
  Patient Health Questionnaire 2 - Scores range from 0-6. Higher scores above 3 indicates that major depressive disorder is likely.
  Patient Health Questionnaire 9 - Scores range from 0-27. Higher scores indicates that major depressive disorder is likely.
Post-traumatic Stress Disorder | Baseline, an average of 5 months after the start of the intervention, and immediately after the intervention, an average of 10 months
  Diagnostic and Statistical Manual 5 PTSD Checklist - Scores range from 0-80 where higher scores indicate more severe PTSD symptoms
Primary Care Visits | Immediately after the intervention, an average of 10 months
  Healthcare Utilization - Number of primary care visits
Anxiety | Baseline, an average of 5 months after the start of the intervention, and immediately after the intervention, an average of 10 months
  Generalized Anxiety Disorder 7 - Scores range from 0-21, where higher scores indicate more severe anxiety
Behavioral Health Visits | Immediately after the intervention, an average of 10 months
  Number of Behavioral Health Visits
Quality of Behavioral Health Visits | Immediately after the intervention, an average of 10 months
  Description of the quality of any behavioral health visits
Acute Hospital Stays | Immediately after the intervention, an average of 10 months
  Number of acute hospitalizations
Emergency Department Stays | Immediately after the intervention, an average of 10 months
  Number of emergency department visits

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sanchez, PhD, LCSW, Principal Investigator — Baylor Scott and White Health; Ann Marie Warren, PhD, ABPP-RP, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor Scott and White Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller B, Burgos A. Enhancing the Capacity of the Mental Health and Addiction Workforce: A Framework. 2021. www.scattergoodfoundation.org
- [Background] Naslund JA, Tugnawat D, Anand A, Cooper Z, Dimidjian S, Fairburn CG, Hollon SD, Joshi U, Khan A, Lu C, Mitchell LM, Muke S, Nadkarni A, Ramaswamy R, Restivo JL, Shrivastava R, Singh A, Singla DR, Spiegelman D, Bhan A, Patel V. Digital training for non-specialist health workers to deliver a brief psychological treatment for depression in India: Protocol for a three-arm randomized controlled trial. Contemp Clin Trials. 2021 Mar;102:106267. doi: 10.1016/j.cct.2021.106267. Epub 2021 Jan 6. PMID 33421650
- [Background] Ma A, Sanchez A, Ma M. The Impact of Patient-Provider Race/Ethnicity Concordance on Provider Visits: Updated Evidence from the Medical Expenditure Panel Survey. J Racial Ethn Health Disparities. 2019 Oct;6(5):1011-1020. doi: 10.1007/s40615-019-00602-y. Epub 2019 Jun 24. PMID 31236800
- [Background] Chao PJ, Steffen JJ, Heiby EM. The effects of working alliance and client-clinician ethnic match on recovery status. Community Ment Health J. 2012 Feb;48(1):91-7. doi: 10.1007/s10597-011-9423-8. Epub 2011 Jun 17. PMID 21681459
- [Background] Hoge MA, Stuart GW, Morris J, Flaherty MT, Paris M Jr, Goplerud E. Mental health and addiction workforce development: federal leadership is needed to address the growing crisis. Health Aff (Millwood). 2013 Nov;32(11):2005-12. doi: 10.1377/hlthaff.2013.0541. PMID 24191093